CLINICAL TRIAL: NCT01158859
Title: Effect of Preoperative Pregabalin on Propofol Induction Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Etienne de Medicis, MD, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRC09-014
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Anesthesia, General; Laparoscopic Surgery
Keywords: Anesthesia, General; Propofol; Pregabalin; Preoperative care; Laparoscopic surgery
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Preoperative administration of pregabalin vs placebo 1 hour before surgery
  Other Names: Lyrica

SUMMARY:
The primary issue is to determine whether preoperatively administered pregabalin decreases the necessary dose of propofol during induction of general anesthesia. The investigators secondary issue is to test if preoperatively administered pregabalin decreases anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic gynaecologic surgery
* Age 18-40 years
* ASA class I or II
* Body mass index 18-30

Exclusion Criteria:

* Allergic to pregabalin or gabapentin
* Chronic renal failure
* Alcohol or drug abuse
* Chronic analgesic use other than acetaminophen or NSAID
* Already taking gabapentin, pregabalin, benzodiazepin or antidepression drug
* Known neurological deficiency
* Suspected difficult intubation or ventilation
* Atypical pseudocholinesterases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Propofol induction dose | 1 hour
  Evaluation of the hpreoperative pregabalin Vs placebo effect on propofol induction dose needed to induce general anesthesia assessed by entropy in gynaecologic patients undertaking minor surgical procedure.

SECONDARY OUTCOMES:
Preoperative anxiety | 1 hour
  Evaluation of the effect of pregabalin Vs placebo on preoperative anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Etienne de Medicis, MD MSc FRCPC, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Background] Gajraj NM. Pregabalin: its pharmacology and use in pain management. Anesth Analg. 2007 Dec;105(6):1805-15. doi: 10.1213/01.ane.0000287643.13410.5e. PMID 18042886
- [Background] Gilron I. Gabapentin and pregabalin for chronic neuropathic and early postsurgical pain: current evidence and future directions. Curr Opin Anaesthesiol. 2007 Oct;20(5):456-72. doi: 10.1097/ACO.0b013e3282effaa7. PMID 17873599
- [Background] Sills GJ. The mechanisms of action of gabapentin and pregabalin. Curr Opin Pharmacol. 2006 Feb;6(1):108-13. doi: 10.1016/j.coph.2005.11.003. Epub 2005 Dec 22. PMID 16376147
- [Background] Kavoussi R. Pregabalin: From molecule to medicine. Eur Neuropsychopharmacol. 2006 Jul;16 Suppl 2:S128-33. doi: 10.1016/j.euroneuro.2006.04.005. Epub 2006 Jun 9. PMID 16765030
- [Background] Hill CM, Balkenohl M, Thomas DW, Walker R, Mathe H, Murray G. Pregabalin in patients with postoperative dental pain. Eur J Pain. 2001;5(2):119-24. doi: 10.1053/eujp.2001.0235. PMID 11465977
- [Background] Mathiesen O, Jacobsen LS, Holm HE, Randall S, Adamiec-Malmstroem L, Graungaard BK, Holst PE, Hilsted KL, Dahl JB. Pregabalin and dexamethasone for postoperative pain control: a randomized controlled study in hip arthroplasty. Br J Anaesth. 2008 Oct;101(4):535-41. doi: 10.1093/bja/aen215. Epub 2008 Jul 23. PMID 18653493
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. Premedication with pregabalin 75 or 150 mg with ibuprofen to control pain after day-case gynaecological laparoscopic surgery. Br J Anaesth. 2008 Jun;100(6):834-40. doi: 10.1093/bja/aen098. Epub 2008 Apr 29. PMID 18448418
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. A randomized controlled trial of perioperative administration of pregabalin for pain after laparoscopic hysterectomy. Pain. 2008 Jan;134(1-2):106-12. doi: 10.1016/j.pain.2007.04.002. Epub 2007 May 15. PMID 17507163
- [Background] Paech MJ, Goy R, Chua S, Scott K, Christmas T, Doherty DA. A randomized, placebo-controlled trial of preoperative oral pregabalin for postoperative pain relief after minor gynecological surgery. Anesth Analg. 2007 Nov;105(5):1449-53, table of contents. doi: 10.1213/01.ane.0000286227.13306.d7. PMID 17959981
- [Background] Kong VK, Irwin MG. Gabapentin: a multimodal perioperative drug? Br J Anaesth. 2007 Dec;99(6):775-86. doi: 10.1093/bja/aem316. PMID 18006529
- [Background] Memis D, Turan A, Karamanlioglu B, Seker S, Ture M. Gabapentin reduces cardiovascular responses to laryngoscopy and tracheal intubation. Eur J Anaesthesiol. 2006 Aug;23(8):686-90. doi: 10.1017/S0265021506000500. PMID 16805934
- [Background] Fassoulaki A, Melemeni A, Paraskeva A, Petropoulos G. Gabapentin attenuates the pressor response to direct laryngoscopy and tracheal intubation. Br J Anaesth. 2006 Jun;96(6):769-73. doi: 10.1093/bja/ael076. Epub 2006 Apr 4. PMID 16595614
- [Background] Menigaux C, Adam F, Guignard B, Sessler DI, Chauvin M. Preoperative gabapentin decreases anxiety and improves early functional recovery from knee surgery. Anesth Analg. 2005 May;100(5):1394-1399. doi: 10.1213/01.ANE.0000152010.74739.B8. PMID 15845693
- [Background] Johansen JW. Update on bispectral index monitoring. Best Pract Res Clin Anaesthesiol. 2006 Mar;20(1):81-99. doi: 10.1016/j.bpa.2005.08.004. PMID 16634416
- [Background] Bein B. Entropy. Best Pract Res Clin Anaesthesiol. 2006 Mar;20(1):101-9. doi: 10.1016/j.bpa.2005.07.009. PMID 16634417
- [Background] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656
- [Derived] Moreau-Bussiere F, Gaulin J, Gagnon V, Sansoucy Y, de Medicis E. Preoperative pregabalin does not reduce propofol ED(50): a randomized controlled trial. Can J Anaesth. 2013 Apr;60(4):364-9. doi: 10.1007/s12630-013-9885-y. Epub 2013 Jan 19. PMID 23334782